CLINICAL TRIAL: NCT06540417
Title: Study of the Neuroprotection and Rehabilitation Promotion of the Non-invasive Trigeminal Nerve Stimulation on Ischemic Stroke Patients
Brief Title: Study of the Effects of the Non-invasive Trigeminal Nerve Stimulation on Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xidian University (Other)
Responsible Party: Principal Investigator, Wei Qin, Professor, Xidian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20231210
Record Dates: First submitted 2024-07-24; First posted 2024-08-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTNS treatment (Active Comparator): Bilateral supraorbital regions were selected as the stimulation sites for external trigeminal nerve stimulation (eTNS).
  Interventions: Device: External trigeminal nerve stimulation
- Control treatment (No Intervention): The standard treatment group received physician-directed treatment for acute ischemic stroke, which included medication and rehabilitation therapy.

INTERVENTIONS:
Device: External trigeminal nerve stimulation — The stimulation parameters were set to 120Hz, 250μs, 30s ON-30s OFF, with the intensity adjusted for patient comfort.
  Arms: eTNS treatment

SUMMARY:
In patients with ischemic stroke, the primary focus revolves around enhancing the neuroprotective and rehabilitative effects of external trigeminal nerve stimulation (eTNS) and elucidating its underlying central mechanisms. Through clinical trials and neuroimaging studies, this research endeavors to 1) investigate the clinical impact of TNS on brain protection and 2) rehabilitation acceleration in ischemic stroke patients, while concurrently exploring the potential central nervous mechanisms involved. The ultimate aim is to contribute a novel therapeutic approach to the clinical management of acute ischemic stroke.

DETAILED DESCRIPTION:
This study conducted a randomized controlled clinical trial with an intention to enroll 60 patients. Patients were randomly assigned in a 1:1 ratio to two groups: 1) External trigeminal nerve stimulation (eTNS) group (intervention group); 2) Standard treatment group (control group). eTNS was administered once daily for 30 consecutive days during the treatment period. The eTNS stimulation protocol entailed targeting the bilateral supraorbital region as the non-invasive stimulation site, with treatment administered for 30 days (once daily, during nighttime sleep for a minimum of 8 hours per day; stimulation parameters set at 120 Hz, 250 μs, 30s ON-30s OFF, with intensity adjusted to individual comfort levels). For the standard treatment group, a series of interventions excluding eTNS, as directed by the treating physician, were administered (including but not limited to medications and rehabilitation therapies). Blood samples and medical history information were collected at baseline. Imaging data were acquired from participants at baseline and 5 days post-treatment. Modified Rankin Scale (mRS), National Institutes of Health Stroke Scale (NIHSS), and Barthel Index (BI) were assessed at baseline, 5 days post-treatment, at the end of treatment, and at 1- and 2-month follow-ups. Additionally, the 9-item Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder 7-item scale (GAD-7), and Insomnia Severity Index (ISI) were administered at baseline, the end of treatment, and at 1- and 2-month follow-ups to evaluate participants' emotional well-being and sleep patterns. The recruited sample size met statistical requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Medically diagnosed with acute ischemic stroke;
* Ability to receive trigeminal nerve stimulation within 72 hours post-stroke onset;
* NIHSS (National Institutes of Health Stroke Scale) score ≥ 4;
* Signed informed consent form;
* Ability and willingness to comply with the study requirements.

Exclusion Criteria:

* History of ischemic or hemorrhagic stroke within the past 3 months;
* Patients in a comatose state;
* Severe allergic reaction to MR contrast agents or renal impairment, eGFR <30 ml/min, excluding the use of contrast agents;
* Pregnant or breastfeeding women;
* Any other life-threatening or severe medical condition that may interfere with the completion of the study protocol, including the 3-month follow-up;
* Exclusion from trigeminal nerve stimulation: patients with trigeminal neuralgia or facial pain;
* Current or recent participation in other neuromodulation stimulation therapies within the past 3 months;
* Refusal to sign the informed consent form;
* Presence of contraindications related to MRI scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Response rate after five days of treatment | NIHSS will be assessed five times within 90 days: at baseline (prior to participant enrollment), and on days 5, 30, 60, and 90 post-enrollment.
  The National Institutes of Health Stroke Scale (NIHSS) is employed to evaluate the extent of functional impairment caused by stroke. Comprising 11 test items, the scale's scoring ranges from 0 to 42. Higher scores are indicative of more severe strokes and are positively correlated with the volume of cerebral damage caused by the stroke.
  Response is defined as a decrease in NIHSS (National Institutes of Health Stroke Scale) score by 4 points or more, or a decrease to 0-1 points after treatment. The response rate is the proportion of participants whose NIHSS scores decrease by 4 points or more, or to 0-1 points, compared to baseline.

SECONDARY OUTCOMES:
Infarct volume growth rate | Imaging data will be collected twice within 90 days: at baseline (prior to participant enrollment) and on the fifth day of treatment.
  Defined as the difference in infarct volume on day 5 compared to baseline, divided by the baseline infarct volume.
Change in NIHSS scores | NIHSS will be assessed five times within 90 days: at baseline (prior to participant enrollment), and on days 5, 30, 60, and 90 post-enrollment.
  The National Institutes of Health Stroke Scale (NIHSS) is employed to evaluate the extent of functional impairment caused by stroke. Comprising 11 test items, the scale's scoring ranges from 0 to 42. Higher scores are indicative of more severe strokes and are positively correlated with the volume of cerebral damage caused by the stroke.
  The change in NIHSS score will be determined by subtracting the baseline score from the score at each subsequent time point.
Change in mRS scores | mRS will be assessed five times within 90 days: at baseline (prior to participant enrollment), and on days 5, 30, 60, and 90 post-enrollment.
  The Modified Rankin Scale (mRS) is employed to assess the status of neurological function recovery in stroke patients. This scale is categorized into seven levels with a scoring range from 0 to 6. Each level corresponds to a specific score; higher scores indicate a poorer prognosis, with a score of 6 signifying death.
  The change in mRS score will be calculated by subtracting the baseline score from the score at each subsequent time point.
Change in BI scores | BI will be assessed five times within 90 days: at baseline (prior to participant enrollment), and on days 5, 30, 60, and 90 post-enrollment.
  The Barthel Index (BI) measures the ability of patients to perform daily living activities. Scores range from 0 to 100, with higher scores reflecting greater independence and less dependency.
  The change in BI score will be calculated by subtracting the baseline score from the score at each subsequent time point.
Change in PHQ-9 scores | PHQ-9 will be assessed four times within 90 days: at baseline (prior to participant enrollment), and on days 30, 60, and 90 post-enrollment.
  The Patient Health Questionnaire-9 (PHQ-9) encompasses nine items, each representing a different facet of depressive symptoms. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
  The change in PHQ-9 score will be determined by subtracting the baseline score from the score at each subsequent time point.
Change in GAD-7 scores | GAD-7 will be assessed four times within 90 days: at baseline (prior to participant enrollment), and on days 30, 60, and 90 post-enrollment.
  The Generalized Anxiety Disorder Scale (GAD-7) is used to assess the emotional state of patients. The Generalized Anxiety Disorder Scale (GAD-7) comprises seven items, with a total possible score ranging from 0 to 21. An elevated score suggests a more pronounced level of anxiety.
  The change in GAD-7 score will be determined by subtracting the baseline score from the score at each subsequent time point.
Change in ISI scores | ISI will be assessed four times within 90 days: at baseline (prior to participant enrollment), and on days 30, 60, and 90 post-enrollment.
  The Insomnia Severity Index （ISI） is utilized to assess the severity of insomnia and its impact on physical health, daily function, and quality of life. This scale includes seven items, with a total scoring range from 0 to 28. Higher scores denote more severe insomnia.
  The change in ISI score will be determined by subtracting the baseline score from the score at each subsequent time point.
Correlation Between Time to Treatment and Intervention Outcomes | The time from stroke onset to treatment will be recorded prior to enrollment.
  The correlation between the hours from stroke onset to treatment and intervention outcomes (defined by NIHSS score improvement or no improvement) will be assessed.
Correlation Between Blood Inflammatory Markers and Stroke Severity and Intervention Outcomes | Blood samples will be collected at baseline (prior to participant enrollment)
  Blood samples will be collected at baseline (prior to participant enrollment) to measure levels of TNF-α and IL-6 (pg/ml). The correlation between these levels and intervention outcomes (defined by NIHSS score improvement or no improvement) will be analyzed.
Correlation Between Medical History and Intervention Outcomes | Medical History will be collected at baseline (prior to participant enrollment)
  Participants' medical history, including diabetes, hypertension, coronary artery disease, and history of cerebral infarction, will be collected at baseline to examine the relationship between medical history and the efficacy of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Zhao, Doctor, Principal Investigator — Shaanxi Provincial People's Hospital; Wei Qin, Phd, Principal Investigator — Xidian University
Locations (1):
- Xidian University, Xi'an, Shaanxi, China